CLINICAL TRIAL: NCT00968240
Title: Phase I Trial of Super-Selective Intraarterial Intracranial Infusion of Avastin (Bevacizumab) For Treatment of Relapsed/Refractory Glioblastoma Multiforme and Anaplastic Astrocytoma
Brief Title: Super-Selective Intraarterial Intracranial Infusion of Avastin (Bevacizumab)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, John A. Boockvar, Associate Professor, Northwell Health
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0901010185
Record Dates: First submitted 2009-08-26; First posted 2009-08-28 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Glioblastoma Multiforme; Anaplastic Astrocytoma
Keywords: GBM; AA; AO; Brain; Tumors; Malignant; Glioblastoma; Multiforme; Anaplastic; Astrocytoma
MeSH Terms: conditions — Glioblastoma; Astrocytoma; Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Super-Selective Intraarterial Intracranial Infusion of BEVACIZUMAB — This phase I clinical research trial will test the hypothesis that Bevacizumab can be safely used by direct intracranial superselective intraarterial infusion up to a dose of 10mg/kg to ultimately enhance survival of patients with relapsed/refractory GBM/AA.
  Day 0: Intraarterial Avastin single dose (starting at 2mg/kg and up to 10mg/kg) after Mannitol to open the blood brain barrier.
  Other Names: Avastin

SUMMARY:
The high-grade malignant brain tumors, glioblastoma multiforme (GBM) and anaplastic astrocytoma (AA), comprise the majority of all primary brain tumors in adults. This group of tumors also exhibits the most aggressive behavior, resulting in median overall survival durations of only 9-12 months for GBM, and 3-4 years for AA. Initial therapy consists of either surgical resection, external beam radiation or both. All patients experience a recurrence after first-line therapy, so improvements in both first-line and salvage therapy are critical to enhancing quality-of-life and prolonging survival. It is unknown if currently used intravenous (IV) therapies even cross the blood brain barrier (BBB). Superselective Intraarterial Cerebral Infusion (SIACI) is a technique that can effectively increase the concentration of drug delivered to the brain while sparing the body of systemic side effects. One currently used drug called, Bevacizumab (Avastin) has been shown to be active in human brain tumors but its actual CNS penetration is unknown. This phase I clinical research trial will test the hypothesis that Bevacizumab can be safely used by direct intracranial superselective intraarterial infusion up to a dose of 10mg/kg to ultimately enhance survival of patients with relapsed/refractory GBM/AA. By achieving the aims of this study we will determine the toxicity profile and maximum tolerated dose (MTD of SIACI Bevacizumab. We expect that this project will provide important information regarding the utility of SIACI Bevacizumab therapy for malignant glioma, and may alter the way these drugs are delivered to our patients in the near future.

DETAILED DESCRIPTION:
The current standard of care for recurring GBM is for patients to receive Bevacizumab (Avastin) intravenously (IV) at 10mg/kg with CPT-11 (Irinotecan) every two weeks until their tumor grows more than 25%. At that point, these patients are deemed treatment failures and are given another treatment. Because of the blood brain barrier (BBB) where IV drugs do not penetrate the blood vessel walls well to get into the brain, no one knows for sure if these IV drugs actually get into the brain after infusion. Previous studies have shown that if you want to increase your penetration of drug to the brain, that intra-carotid artery (intraarterial) delivery is superior to standard intravenous delivery. Previous techniques using intra arterial (intracarotid) infusion still were non-selective as drug delivery still went to all blood vessels in the brain, so patients still had significant adverse events, such as blindness. Newer techniques in interventional neuroradiology have allowed for a more selective delivery of catheters higher up into the arterial tree where agents such as chemotherapies, can be delivered without the risk of adverse affects such as blindness. In fact, studies here at Cornell and MSKCC have developed very new and exciting super selective intraarterial delivery treatment for Pediatric Eye Tumors with little toxicity. Therefore, this trial will ask one simple question: Is it safe to delivery a patient's first dose of Avastin intraarterially using these super selective delivery techniques instead of the standard intravenous route of administration? This should not only increase the amount of drug that gets to the tumor but also spare the patient any adverse effects from a less selective delivery. During that single dose of intraarterial Avastin, the patient will also receive a dose of mannitol that opens up the blood brain barrier to improve delivery of the agent to the brain. After that single dose of Mannitol and Avastin intraarterially, the patient will be evaluated for 4 weeks to assess for toxicity. If no toxicity, then the patient will go on and get the standard chemotherapy (Avastin and CPT-11) every two weeks as is routine unless they fail. After this you are done with the "experimental" aspects of the protocol. This is a Phase I trial that is designed to test the safety of the single dose intraarterial delivery of Avastin and Mannitol, prior to starting standard IV Avastin and CPT-11.

In summary:

Current Standard of Care:

Day 0: Intravenous Avastin (10mg/kg) and CPT-11 Day 14, 28 (and every two weeks thereafter): Intravenous Avastin and CPT-11

Experimental portion of this proposal:

Day 0: Intraarterial Avastin single dose (starting at 2mg/kg and up to 10mg/kg) after Mannitol to open the blood brain barrier Day 28 (and every two weeks thereafter): Intravenous Avastin and CPT-11

1. Subjects will first be treated with Mannitol prior to chemotherapy infusion (Mannitol 25%; 3-10 mL/s for 30seconds) in order to disrupt the blood brain barrier. This technique has been used in several thousand patients in previous studies for the IA delivery of chemotherapy for malignant glioma.
2. To add a single intraarterial delivery (SIACI) of the Avastin prior to beginning the standard IV Avastin and CPT-11 therapy for patients with recurring or relapsing high grade glioma. After a one cycle observation period assess for toxicity from the IA infusion, the subject will receive Intravenous (IV) bevacizumab 10 mg/kg and irinotecan (CPT-11) 125mg/m2 every 14 days as is standard therapy for relapsing recurring GBM.

The dose escalation algorithm is as follows: We will use a single intracranial superselective intraarterial infusion of Avastin, starting at a dose of 2mg/kg in the first three patients. Assuming no dose limiting toxicity during the first 28 days after IA infusion, the patient will then begin their standard chemotherapy regimen which is Avastin and CPT-11 every two weeks. The doses will be escalated to 4,6,8 and finally 10mg/kg in this Phase I trial.

Inclusion criteria Include: Males or females, ≥18 years of age, with documented histologic diagnosis of relapsed or refractory glioblastoma multiforme (GBM), anaplastic astrocytoma (AA) or anaplastic mixed oligoastrocytoma (AOA).

Both hematologic and non-hematologic toxicity will be determined and scored according to the NCI Common Toxicity Criteria (version 3.0). Monitoring will be conducted by post procedure CT scan (at 6-12 hours post procedure), serial history, neurological and physical examinations together with serial blood counts, prothrombin time (PT), partial thromboplastin time (PTT) and chemistries. MRI will be performed every two cycles or approximately every two months.

Response will be evaluated after two cycles of chemotherapy via a MRI with the injection of contrast. Subjects who show an objective response (reduction in tumor size) or stable disease after 2 cycles of treatment will be able to continue on study. Progressive disease will require that subjects be taken off the research protocol. The following will be evaluated every cycle, and then during follow-up: neurological examination, physical examination, performance status, laboratory parameters and review of adverse reactions. Contrast enhanced MRI (MRI with gadolinium is the preferable imaging study except in case where MRI is contraindicated i.e., in those with pacemakers or metallic implants. In these subjects, CT with contrast is acceptable) will be performed every two-treatment cycles under this research protocol. The following subjects will be taken off protocol: those with progressive disease; those who experience dose-limiting toxicity (DLT). Follow-up will continue until disease progression or death. Survival will be measured from the time of the first dose of IA Avastin® (given at the start of each treatment cycle).

The patient will not be responsible for any additional costs associated with enrollment in the trial. All costs of the IA delivery will be submitted to the patient's insurance provider. WCMC will not be named as a sponsor of the study nor will it cover the cost of the experimental procedure.

ELIGIBILITY:
INCLUSION

* Male or female patients of greater or equal18 years of age.
* Patients with a documented histologic diagnosis of relapsed or refractory glioblastoma multiforme (GBM), anaplastic astrocytoma (AA)
* Patients with a histologically confirmed low-grade brain tumor who relapse with an enhancing tumor on MRI can be evaluated for toxicity only.
* Patients must have at least one confirmed and evaluable tumor site.

  *A confirmed tumor site is one in which is biopsy-proven. NOTE: Radiographic procedures (e.g., Gd-enhanced MRI or CT scans) documenting existing lesions must have been performed within three weeks of treatment on this research study.
* Patients must have a Karnofsky performance status greater or equal to 60% (or the equivalent ECOG level of 0-2) (see Appendix A; Performance Status Evaluation) and an expected survival of greater or equal to three months.
* Patients must be able to understand informed consent. Informed consent must be obtained at the time of patient screening.
* Because of known concerns with Avastin and wound healing, all craniotomy patients are eligible for the treatment if they have had a craniotomy > two weeks prior to IA therapy. Craniotomy after SIACI bevacizumab therapy should wait 4 weeks.
* Pre-enrollment coagulation parameters (PT and PTT) must be less than or equal to1.5X the IUNL.
* Patients must have adequate hematologic reserve with WBC greater than or equal to 2800/mm3, absolute neutrophils greater than or equal to1500/mm3 and platelets greater than or equal to 100,000/ mm3.
* Pre-enrollment chemistry parameters must show: bilirubin<1.5X the institutional upper limit of normal (IUNL); AST or ALT<2.5X IUNL and creatinine<1.5X IUNL.
* No external beam radiation for four weeks prior to treatment under this research protocol.
* No chemotherapy for three weeks prior to treatment under this research protocol.

EXCLUSION:

* Patients previously treated with more than 6 cycles (28 days each) of Bevacizumab at 10/mg/kg.
* Women who are pregnant or lactating.
* Women of childbearing potential and fertile men who decline to use effective contraception during and for a period of three months after the treatment period.
* Patients with significant intercurrent medical or psychiatric conditions that would place them at increased risk or affect their ability to receive or comply with treatment or post-treatment clinical monitoring.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
To determine the safety of superselective intracranial intraarterial infusion of Avastin up to a dose of 10mg/kg IA. | 3 years

SECONDARY OUTCOMES:
Composite overall response rate: The composite overall response rate (CORR) will be examined. The overall response proportion along with a 95% confidence interval will be estimated via binomial proportions. | 3 years
Six-month progression-free survival (PFS) and overall survival (OS) will be assessed by Kaplan-Meier survival analysis, assuming adequate follow-up time. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: John Boockvar, MD, Principal Investigator — Weill Cornell Medical College-New York Presbyterian Hospital
Locations (1):
- Lenox Hill Brain Tumor Center, New York, New York, United States